CLINICAL TRIAL: NCT06774755
Title: Reconstructions of Chest Wall Defects: a Retrospective Study
Acronym: PLAST-CHEST
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PLAST-CHEST
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Chest Wall Deformity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients requiring thoracic reconstruction often suffer from numerous comorbidities, such as obesity, diabetes, atherosclerosis and cardiovascular diseases, respiratory diseases. The clinical picture of these patients must be carefully stabilized in the preoperative period since the listed diseases are associated with a poor reconstructive outcome. Furthermore, it is necessary to preoperatively determine the spirometric characteristics in cases where the intervention may alter the respiratory dynamics to evaluate the patient's ability to tolerate the procedure. The primary objective of the study is to identify the best diagnostic-therapeutic approach in cases of complex chest wall defects, retrospectively evaluating the outcomes and therapeutic choices implemented, through a reassessment of the interventions performed and the clinical progress of patients undergoing complex thoracic and sternal reconstruction interventions managed in a multidisciplinary and non-multidisciplinary manner

DETAILED DESCRIPTION:
Currently there are no univocal universally accepted guidelines regarding the intervention to be performed in case of complex chest wall reconstructions or for the treatment of sternal wound dehiscences. Different options are described, both for the demolition phase and for the reconstructive phase in the thoracic and sternal area. The choice of one method rather than the other is currently largely based on the experience and preference of the specific working group. The importance of the study lies in the attempt to analyze the choices made in the diagnostic and therapeutic phase (demolitive, reconstructive, pharmacological) on patients treated at the AOU Sant'Orsola (now IRCCS) in past years. The secondary objective of the study is to improve the multidisciplinary management of patients who are candidates for complex chest reconstructions.

In particular, the drafting of a multidisciplinary therapeutic protocol that uses algorithms to optimize the choice of surgical procedure and medical therapy in terms of resolution of the problem, hospitalization times, and patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing sternal or thoracic reconstruction in collaboration or not with the Reconstructive Plastic Surgery Unit
* Obtaining informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients meeting the inclusion criteria will be counted, starting from January 1, 2010 to January 1, 2023.
  It is estimated that approximately 100 patients will meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Technical Success | From the first patient enrolled, up to the 100th patient
  Thechnical success is evaluated by duration of surgery, complications and need for reoperation, and hospitalization time

CONTACTS AND LOCATIONS:
Overall Officials: Marco Pignatti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS AOU di Bologna Policlinico di Sant'Orsola, Bologna, Italy